CLINICAL TRIAL: NCT07202897
Title: LA-HCM Study : Rivaroxaban for Antithrombotic Prevention in Hypertrophic Cardiomyopathy Patients With Abnormal Left Atrial Strain: A Randomized Multicenter Trial
Brief Title: LA-HCM Study : Rivaroxaban for Antithrombotic Prevention in Hypertrophic Cardiomyopathy Patients With Abnormal Left Atrial Strain.
Acronym: LA-HCM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35RC22_9771_LA-HCM; 2024-511084-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulant treatment Rivaroxaban (Experimental)
  Interventions: Drug: Anticoagulant treatment Rivaroxaban
- Best medical therapy (Active Comparator)
  Interventions: Other: Best medical therapy

INTERVENTIONS:
Drug: Anticoagulant treatment Rivaroxaban — Anticoagulant treatment Rivaroxaban in addition to best medical therapy
  Arms: Anticoagulant treatment Rivaroxaban
Other: Best medical therapy — Best medical therapy alone
  Arms: Best medical therapy

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a common (> 1/500 in the general adult population) genetically transmitted disease impacting markedly patients' lives from the early ages to the latest. The phenotype as the prognosis of HCM may greatly differ from one patient to another: most patients present no or few symptoms and a near-normal lifespan, while others are severely symptomatic. Paroxysmal, persistent or permanent atrial fibrillation (AF) is frequent in HCM, occurring in more than 20%-25% of patients and is often considered as an important turning point for the quality of life of these patients. AF decreases cardiac output and exercise tolerance, increases hospitalization rate, and markedly increase the risk of embolic stroke with the need for life-anticoagulation. It has been shown that stroke may precede AF discovery and that it may occur at young ages with devastation consequences. AF also may trigger sudden cardiac death.

Observational studies have been conducted to search for parameters which correlate with the risk of AF (P wave duration and supra-ventricular burst on the Holter-ECG monitoring, L-wave morphology, degree of hypertrophy, clinical parameters-comorbidities, and size of the left atrium) with no real impact on clinical management. Left Atrial strain (LA-strain) has been recently demonstrated relevant (for instance our pilot work (for predicting stroke and/or AF (a cut-off of 15% is highly specific, 20% being the optimal cut-off). LA-strain (cut-off 20%) could be used for defining the patients that might require preventive anticoagulation therapy.

A randomized clinical trial is needed to extend the use of anticoagulation therapy to patients in sinus rhythm but identified to be at risk for AF.

Of note, it has been demonstrated that in this population, stroke occurred in 67% of the patients without any clinical atrial arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

1. 40 - 80 years of age
2. 50 and 120 kg of weight
3. In sinus rhythm
4. Prior confirmed diagnosis of "primary" hypertrophic cardiomyopathy
5. Left Atrial reservoir strain measured ≤20% (corelab confirmation)
6. Signature of an informed consent
7. Highly effective contraceptive methods for women of childbearing potential from at least 14 days prior to start treatment, throughout the study treatment period, and until at least 4 weeks after the last dose of study medication

Exclusion Criteria:

1. Secondary hypertrophic cardiomyopathy (aortic stenosis, hypertension, amyloidosis and all phenocopies…)
2. Signs of heart failure
3. Hospitalization
4. Uncontrolled blood pressure
5. Creatinine clearance <30 mL/min (Cockcroft)
6. Severe liver dysfunction, cirrhosis Child B or C
7. Any anticoagulation therapy in the 15 days prior to enrollment
8. Any cardiac surgery in the 30 days prior to enrollment
9. Documented atrial arrhythmia
10. Any major bleeding in the 90 days prior to enrollment
11. Need to be on dual antiplatelet therapy (aspirin >100 mg daily and a P2Y12 inhibitor, i.e. clopidogrel, ticagrelor, prasugrel…).
12. Contraindication for a brain magnetic resonance imaging exam
13. Known hypersensitivity or others contraindications to Rivaroxaban (refer to contraindications)
14. Ischemic stroke or intracranial hemorrhage in the 30 days prior to enrollment
15. Active endocarditis at the time of enrollment
16. Concomitant combined strong P-gp and CYP3A4 inducers or inhibitors
17. Active cancer or life expectancy less than 3 years
18. Non-compliant
19. Participation in another interventional clinical trial
20. Protected person (adults legally protected (under judicial protection, guardianship or supervision), person deprived of their liberty, pregnant woman, lactating woman or planning pregnancy during the study period and minor)
21. Absence of coverage by a social security scheme

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
all-cause death, myocardial infarction, stroke and systemic embolism | 2 years

SECONDARY OUTCOMES:
Bleeding | 2 years
  Number of observed bleeding divided by the sum of person-time at risk
Ischemic endpoints and bleeding to estimate the net clinical benefit | 2 years
  The net clinical benefit is calculated by subtracting the rate of excess bleeding events attributable to the experimental arm from the rate of excess ischemic events possibly prevented by the experimental arm
Atrial arrhythmias | 2 years
Left Atrial reservoir strain | 2 years
Kansas City Cardiomyopathy Questionnaire | 2 years
  score between 0 and 100. A high score indicates a better quality of life and a lower score indicates a deterioration in quality of life